CLINICAL TRIAL: NCT06077617
Title: Bedside Ultrasound Assessment of Feeding Tube Position in the Intensive Care Unit: the US-FEED Study
Brief Title: Bedside Ultrasound Assessment of Feeding Tube Position in the Intensive Care Unit
Acronym: US-FEED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0627
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Tube Feeding
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic group: Adult ICU patients submitted to feeding tube placement according to institutional standard operating procedure

SUMMARY:
This diagnostic accuracy study aims to evaluate the performance of bedside ultrasound compared to x-ray in detecting the correct position of feeding tubes among critically ill adult patients. The main questions it aims to answer are: • diagnostic accuracy of bedside ultrasound • feasibility of its wide adoption among practitioners with minimal training in busy intensive care units.

DETAILED DESCRIPTION:
This multicenter diagnostic accuracy study consists of a non-consecutive convenience sample of adult patients admitted to the intensive care unit starting from March 2023 who require a feeding tube as defined by the medical attending team.

Right after feeding tube placement following the institutional standard operating procedure, attending physicians perform bedside ultrasound assessment to verify the correct position of the tube. They report whether or not visualizing the feeding tube in four steps: 1) in the esophagus from either the right or left side of the patient's neck; 2) in the transverse view of the patient's epigastrium; 3) in the longitudinal view of the patient's epigastrium and 4) during the injection of 20 mL of air into the tube to detect the 'fogging sign.' Finally, the abdominal radiograph (gold standard) confirms the gastric or duodenal placement of the feeding tube.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old;
* Need for a tube feeding for receiving diet and/or medication, as indicated by the medical team;
* Blind insertion of a tube feeding in the intensive care unit, following the standard operating procedure;
* Presence of a trained physician for ultrasound scanning of the tube feeding immediately after installation.

Exclusion Criteria:

* Major abdominal postoperative wounds, peritoneostomy, or any other conditions that preclude ultrasound abdominal examination;
* Exclusive presence of a gastric decompression probe, which does not require radiographic confirmation;
* Tube feeding introduced under digestive endoscopy guidance;
* Gestation;
* Abdominal radiography confirming the tube position obtained before the ultrasound assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted in the intensive care unit undergoing a tube feeding placement as defined by the attending medical team and in accordance with the institutional standard operating procedure.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | The expected time between ultrasound assessment and abdominal radiography is under 2 hours..
  Estimating sensitivity, specificity, positive predictive rate, negative predictive rate, and total accuracy of bedside ultrasound compared with abdominal radiography (gold standard). A receiver operating characteristic (ROC) curve will display the discriminatory properties of the ultrasound assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina P Antonio, PhD, Principal Investigator — HCPorto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided